CLINICAL TRIAL: NCT05022745
Title: ERAS Protocol for Single-level Posterior Lumbar Arthrodesis; a Randomized Prospective Study
Brief Title: ERAS Protocol for Single-level Posterior Lumbar Arthrodesisprospective Study.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ Nikolaas (Other)
Responsible Party: Principal Investigator, Erik Van de Kelft, M.D., PhD, Head of neurosurgery department, AZ Nikolaas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERAS for PLIA 2020-12
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Mobility; Opioid Use; Instable Spine
Keywords: Enhanced recovery after surgery (ERAS); Posterior lumbar Interbody arthrodesis (PLIA); length of hospital stay (LOS); opioid use

STUDY DESIGN:
Intervention Model Description: Randomized controlled study in patients undergoing PLIA
Masking Description: The interventions described in the patient information brochure make masking impossible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): Posterior lumbar interbody fusion Multimodal, multidisciplinary patient care.
  Interventions: Other: Multimodal, multidisciplinary approach
- Standard group (Active Comparator): Posterior lumbar interbody fusion Standard treatment pre-, per-, and post-operative
  Interventions: Other: Multimodal, multidisciplinary approach

INTERVENTIONS:
Other: Multimodal, multidisciplinary approach — The patient management is adapted pre-operatively, per-operatively and post-operatively
  Other Names: standard treatment

SUMMARY:
Enhanced Recovery After Surgery (ERAS) is a multidisciplinary, multimodal approach aiming to improve surgical outcomes. This study compares the length of hospital stay of patients undergoing single-level posterior lumbar arthrodesis and treated with the ERAS protocol with the hospital stay of patients treated according to the standard protocol.

DETAILED DESCRIPTION:
Hundred and ten patients scheduled for single-level posterior lumbar arthrodesis (PLIA) will be randomized to be treated by the standard protocol or the Enhanced Recovery After Surgery (ERAS) protocol. The ERAS protocol differs from the standard protocol in 4 phases: pre-operative counseling and intake, day of surgery, the pre-operative patient preparation, the per-operatively used analgesic and anesthetic drug combination, and the post-operative care consisting of a more intensive physical therapy in the ERAS group. It is the objective the mobilize patients more rapidly without compromising the comfort in terms of pain.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a single level PLIA as treatment of mono segmental degenerative instability, as seen on dynamic X-rays, after the failure of 6 months conservative therapy Capable of understanding the provided information Giving informed consent

Exclusion Criteria:

* Revision surgery Arthrodesis for trauma, neoplasms, infection, or listhesis due to lysis. High dose opioid use (step 3 of the WHO pain ladder) Diabetes Cognitive impairment (baseline dementia, cognitive dysfunction, or inability to consent to participate).

Known kidney insufficiency: GFR <30 mL/min/1.73 m2 Allergy/intolerance/contraindication to any medication or component included in the ERAS pathway protocol Patients with a risk factor for reflux

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 2-3 days + 11 days
  Number of days hospitalization

SECONDARY OUTCOMES:
Pain intensity | day of discharge
  pain intensity on the day of discharge, measured on a 11-point numeric rating scale
Analgesic use, including opioids | 2-3
  type and dose of analgesics used
11-days readmission rate | discharge + 11 days
  patients who return to the hospital for reasons linked to the recovery after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Nikolaas, Sint-Niklaas, Belgium

IPD SHARING:
Plan to Share IPD: No